CLINICAL TRIAL: NCT03149783
Title: A Randomized Controlled Trial to Determine if Pre- and Post- Operative Regional Pain Control (Transversus Abdominis Plane Block) With Ropivacaine Versus Placebo Leads to Lower Anesthetic and Narcotic Dosing, and Alters Pain Scores
Brief Title: Study to Determine if Pre- and Post- Operative TAP Catheters With Ropivacaine Versus Placebo Affects Anesthetic, Narcotic Dosing, and Pain Scores
Acronym: TAP RCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-1078
Record Dates: First submitted 2017-03-10; First posted 2017-05-11 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative; Delirium; Anesthesia, Local
MeSH Terms: conditions — Pain, Postoperative; Delirium | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Double Blind Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: "Study drug" label of drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine (Experimental): Participants will have bilateral TAP catheters placed along with continuous infusion of ropivacaine.
  Interventions: Drug: Ropivacaine HCL
- Placebo (Placebo Comparator): Participants will have bilateral TAP catheters placed along with continuous infusion of placebo.
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: Ropivacaine HCL — Ropivacaine injected after placement of catheters, then infused during the operation
  Arms: Ropivacaine
Drug: sodium chloride — Placebo
  Other Names: saline
  Arms: Placebo

SUMMARY:
A randomized controlled trial to determine if pre- and post- operative regional pain control (transversus abdominis plane block) with ropivacaine versus placebo leads to lower anesthetic and narcotic dosing, and alters pain scores.

This study plans to learn more about regional anesthesia and pain control during abdominal surgery. The study will gather data about the effectiveness of continuous catheter infusion of local anesthetic after an abdominal operation. Outcomes include pain scores, IV pain medicine requirements, and delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age >=50 years.
* Subjects will be undergoing an elective intra-abdominal or abdominal wall operation, including pelvic operations. Surgery specialties included are general surgery, surgical oncology, urology, gynecology, plastic surgery.

Exclusion Criteria:

* Subjects with a history of dementia or aphasia, as visual analog scale and confusion assessment will be unreliable.
* Patients with an epidural or spinal catheter block.
* Patients who do not speak English so that a language barrier is not confused with VAS scoring or confusion.
* Patients who are abusing alcohol defined by a high AUDIT score (>8) will be excluded.
* History of bipolar disorder or a psychotic disorder (such as a psychotic major depression, schizophrenia, schizoaffective disorder, or psychosis in Alzheimer's disease or other dementia).
* Patients with a documented allergy to ropivacaine or other sodium channel blockers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | Days 0-7 following the operation
  Pain scores from the visual analog scale

SECONDARY OUTCOMES:
Amount of anesthetic | During the operation
  MAC of inhalational agent, or total amount of IV anesthetic used during the operation
Amount of narcotic administered postoperatively | Days 0-7 postop
  Amount of morphine equivalents per day measured after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Robinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver Veterans Affairs Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No sharing